CLINICAL TRIAL: NCT04351412
Title: Comparison of Dentin Hypersensitivity Reduction Over a 1-month Period Between a Single Topical Application of a Dentin-desensitizing Agent (Gluma) and Other Materials: A Randomized Clinical Trial
Brief Title: Comparison of Dentin Hypersensitivity Reduction Over a 1-month Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Dr.Samar Abuzinadah, Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 129-09-19
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Dentin Sensitivity
Keywords: Gluma; Desensitizing agent; Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity | interventions — Gluma

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tactile stimulus (Active Comparator): The tactile stimulus was examined using an explorer (# 17/23), passing at a right angle to the bucco-cervical tooth surface of concern. Contributors evaluated participants' pain score on a 10-point visual analogue scale (VAS). The stimulus was used to assess dentine hypersensitivity at baseline and immediately after completion of treatment. Subjects were also recalled for re-evaluation at 2 weeks and at 1 month after desensitizing treatment.
  Interventions: Other: Gluma; Other: fluoride varnish; Other: Tetric N-Bond self-etch adhesive
- Air blast stimulus (Active Comparator): For air blast stimuli, air was delivered by a three-way syringe from a typical dental unit air syringe at 40 psi (± 10 psi) and 70 °F (± 5 °F). The air flow was aimed at the tooth surface of concern, for 1 second, from a distance of 1 cm. The air blast stimulus scores were assessed by the Schiff Cold Air Sensitivity Scale 18. DH was assessed for air blast stimuli at baseline and immediately after completion of treatment. Subjects were also recalled for re-evaluation at 2 weeks and at 1 month after desensitizing treatment.
  Interventions: Other: Gluma; Other: fluoride varnish; Other: Tetric N-Bond self-etch adhesive
- Cold stimulus (Active Comparator): For cold hypersensitivity assessment, the tooth was isolated using cotton rolls; then, a few drops of extremely cold water were delivered to the tooth from a syringe that had previously been cooled. The cold stimulus scores were assessed by the Schiff Cold Air Sensitivity Scale 18. DH was assessed for cold stimulus at baseline and immediately after completion of treatment. Subjects were also recalled for re-evaluation at 2 weeks and at 1 month after desensitizing treatment.
  Interventions: Other: Gluma; Other: fluoride varnish; Other: Tetric N-Bond self-etch adhesive

INTERVENTIONS:
Other: Gluma — Gluma is desensitizing agent by (Heraeus Kulzer, Armonk, NY, USA) claimed to treat dentine hypersensitivity in exposed cervical teeth surfaces and was applied to participants using a mini brush applicator tip onto the exposed hypersensitive tooth surface requiring treatment and was allowed to dry for 60 seconds. Then Dentine hypersensitivity (DH) was assessed for tactile, cold, and air blast stimuli immediately after completion of treatment. Subjects were also recalled for re-evaluation at 2 weeks and at 1 month after desensitizing treatment.
Other: fluoride varnish — fluoride varnish is usually applied to patients to prevent caries development but was claimed in some cases to also relief dentine hypersensitivity and was applied as a thin layer to the surface of the tooth using an applicator. The varnish set rapidly, and thereafter moisture contamination was not a concern. Patients were advised to not brush or floss their teeth for a couple of hours and to abstain from hot beverages. DH was assessed for tactile, cold, and air blast stimuli immediately after completion of treatment. Subjects were also recalled for re-evaluation at 2 weeks and at 1 month after desensitizing treatment.
Other: Tetric N-Bond self-etch adhesive — Tetric N-Bond self-etch adhesive is one step dental adhesive and is also claimed to relief dentine hypersensitivity due to blockage of dentinal tubules. It was applied according to the manufacturer's instructions, in a thick layer, for at least 30 seconds, using a light brushing motion. Then, it was dried with a steady stream of air for 3 seconds and light-cured for 10 seconds. DH was assessed for tactile, cold, and air blast stimuli immediately after completion of treatment. Subjects were also recalled for re-evaluation at 2 weeks and at 1 month after desensitizing treatment.

SUMMARY:
Here we assessed the clinical effectiveness of Gluma, fluoride varnish, and the Tetric N-Bond one-step self-etch system in alleviating DH instantly and over 1 month, after a single topical application.A randomized, double-blind, clinical trial was conducted on 55 patients (25 males, 30 females; age: 20-49 years). Seventy teeth were randomly assigned to three groups: Gluma (n = 24); fluoride varnish (n = 23); and Tetric N-Bond adhesive (n = 23). Sensitivity to tactile, air blast, and cold stimuli were investigated.. A visual analogue scale was used to assess tactile stimuli, and the Schiff Cold Scale to assess air blast and cold stimuli. DH was evaluated immediately post-treatment, and at the 2-week and 1-month follow-up. Between-group and within-group comparisons were made.

ELIGIBILITY:
Inclusion Criteria:

* Middle-aged adult population who usually complains of Dentin Hypersensitivity.
* Age range 20-49 years, that visit the dental hospital at King Abdul-Aziz university (KAUDH) who would have at least one or two teeth with DH
* Those with recession of the gingiva, teeth erosion or abrasion.
* Patients agreed to participate in the study.

Exclusion Criteria:

* Patients going through professional desensitizing treatment during the previous three months; Using desensitizing tooth paste in the last two months
* Chronic; far on progress periodontal disease; treatment for periodontal disease;
* Teeth with ICDAS (International Caries Detection and Assessment System) score 4
* Teeth diagnosed for irreversible pulpitis; root canal treated teeth
* Teeth covered with crowns; bridge
* Teeth with cervical restorations interfering with the evaluation
* Medically compromised patients currently using medications like anticonvulsants, antihistamines, antidepressants, sedatives or daily analgesics.
* Pregnant or lactating women; were also excluded.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-02-09 (Actual); Study Completion 2020-02-09 (Actual)

PRIMARY OUTCOMES:
Assess dentine hypersensitivity score to stimuli at Baseline | Baseline before treatment
  Scores of DH for tactile stimulus were recorded using visual analogue scale and for cold, and air blast stimuli using the Schiff Cold Air Sensitivity Scale 18 at baseline.
Assess dentine hypersensitivity score to stimuli immediately after treatment by intervention | From baseline to immediately after treatment with intervention
  Scores of DH for tactile stimulus were recorded using visual analogue scale and for cold, and air blast stimuli using the Schiff Cold Air Sensitivity Scale 18 were recorded immediately after treatment with intervention and compared score to baseline.
Assess dentine hypersensitivity to stimuli at two-weeks follow up after treatment by intervention | From baseline to two-weeks follow up after treatment with intervention
  Scores of DH for tactile stimulus were recorded using visual analogue scale and for cold, and air blast stimuli using the Schiff Cold Air Sensitivity Scale 18 were recorded at two-weeks follow up after treatment with intervention and compared score to baseline and immediate treatment scores.
Assess dentine hypersensitivity to stimuli at one month follow up after treatment by intervention | From baseline to one month follow up after treatment with intervention
  Scores of DH for tactile stimulus were recorded using visual analogue scale and for cold, and air blast stimuli using the Schiff Cold Air Sensitivity Scale 18 were recorded at one month (30 days) follow up after treatment with intervention and compared score to baseline and immediate treatment, and two weeks follow up visit scores.

CONTACTS AND LOCATIONS:
Overall Officials: Samar H Abuzinadah, DScD, Study Chair — Assistant Professor, Department of Restorative Dentistry, King Abdul-Aziz University, Jeddah, Saudi Arabia; Abdulrahman J Alhaddad, DScD, Study Director — Assistant Professor, Department of Oral and Maxillofacial Prosthodontics, King Abdul-Aziz University, Jeddah, Saudi Arabia
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abuzinadah SH, Alhaddad AJ. A randomized clinical trial of dentin hypersensitivity reduction over one month after a single topical application of comparable materials. Sci Rep. 2021 Mar 24;11(1):6793. doi: 10.1038/s41598-021-86258-3. PMID 33762645